CLINICAL TRIAL: NCT02712892
Title: IntraCranial ANeurysms: From Familial Forms to Pathophysiological Mechanisms
Brief Title: I-CAN Biocollection
Acronym: I-CAN
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC15_0304
Record Dates: First submitted 2016-02-23; First posted 2016-03-18 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For one patient included:
  * 2 Ethylenediaminetetraacetic acid (EDTA) tubes for DNA (5mL)
  * 2 dry tubes for serum (5mL)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Non Interventional Study

SUMMARY:
Intracranial aneurysm (IA) is an asymptomatic cerebrovascular abnormality affecting 3.2% of the general population. The devastating complication of IA is its rupture, resulting in subarachnoid haemorrhage that can lead to severe disability and death. Unfortunately, there are neither reliable clues nor diagnostic tools to predict the formation and/or the fate of an IA in a given individual. Also, there is no pharmacological drug available to prevent the rupture of aneurysm and subsequent subarachnoid haemorrhage. Current treatments are invasive with a significant risk of procedural morbidity. Thus, still now, the management of patients with IA remains extremely challenging and still controversial. Although the pathogenesis of IA has been the subject of many studies for the last decade, the mechanisms underlying IA formation, growth and rupture are still mostly unknown and relevant animal models of IA are not available. Familial history of IA predisposes to IA formation and rupture and increasing evidence suggest a genetic component of IA formation, with heterogeneous modes of inheritance and penetrance. This project, gathering neuroradiologists, geneticists and vascular biologists, addresses the urgent need to understand the pathogenic mechanisms of IA to develop diagnostic and predictive tools of risk of IA. The investigators propose to identify IA-causing variants by whole-exome sequencing in familial forms of the disease. The investigators hypothesises that the functional analysis of the causal/susceptibility variants thus identified will provide clues to understanding the pathological mechanisms of IA formation, and the bases for developing diagnostic tools. This project aims at meeting this challenge. Based on preliminary data that already allowed to identify such a variant, and the combination of genetic and functional investigations, the specific objectives of this project are: - To identify IA-causing variants in familial forms of the disease by whole-exome sequencing; - To understand the function of these genes/variants in the formation and rupture of IA by molecular and cellular approaches and generation of relevant animal models; - To discover potential biomarkers of risk of IA formation and/or rupture.

ELIGIBILITY:
Inclusion criteria indexes and related cases (familial) of intracranial aneurysms:

* Index: Any patient consulting for a major IA and some typical bifurcation with at least one other case reached akin IA 1st degree
* Related: All similar to the first degree, aged 20 or more, patients with a family background of IA and some typical bifurcation (≥2 achieved) For the latter, directed by screening with Magnetic resonance imaging (MRI) sequence Time of Flight (TOF), axial T2, EGT2.
* biocollection of Written Consent for participation in the collection of biological samples

Inclusion criteria sporadic cases of IA:

* Any patient consulting for IA and some typical bifurcation
* Patients aged 20 years or older
* biocollection of Written Consent for participation in the collection of biological samples

Non Inclusion Criteria:

* Patients who have shown the inability or refusal to sign the consent informed biocollection
* syndromic diagnosis known as AIC provider

  * Marfan Syndrome
  * AOS with SMAD 3
  * Danlos Syndrome Elhers type II and IV
  * Autosomal Dominant Polycystic
  * Moyamoya Syndrome
* character of IA:

  * Dissecting or fusiform
  * Combined with an arteriovenous malformation
  * Blister-like
  * mycotic
* Pathology of the cerebral white matter detected on MRI suggestive:

  * Mutation COL4A1

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The initial stage of this biocollection based on the recruitment of large families for genetic linkage analysis. This is a first step to identify patients with intracranial aneurysms occurring in a family context, and to conduct a comprehensive investigation according to clinical guidelines in force to assess the potentially informative family and ensure their adherence to the prior biocollection. The next step is the fine and accurate phenotyping of each of the family members (imaging) and the collection of a blood sample for DNA extraction for molecular genetic analysis.
  The population recruited will be composed of index and their healthy relatives and cases with sporadic cases and IA. The kinship links will be established from family trees.
Sampling Method: Non-Probability Sample
Enrollment: 3078 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Presence or absence of genetic abnormalitie | Until one year
  Identification of genetic abnormalities segregant with the presence of intracranial aneurysms in the informative families recruited. Sequencing of the whole exome in a cohort of patients carriers of familial forms of intracranial aneurysms.
  Analysis of blood level of the GAIA 1 protein in a large cohort of familial and sporadic carriers of intracranial aneurysms

CONTACTS AND LOCATIONS:
Overall Officials: Hubert DESAL, Pr, Principal Investigator — Nantes University Hospital
Locations (20):
- France (20):
  - Angers University Hospital, Angers
  - Besançon University Hospital, Besançon
  - Bordeaux University Hospital, Bordeaux
  - Henri Mondor Hospital (AP-HP), Créteil
  - Dijon University Hospital, Dijon
  - Grenoble University Hospital, Grenoble
  - La Reunion University Hospital, La Réunion
  - Kremlin-Bicêtre University Hospital (AP-HP), Le Kremlin-Bicêtre
  - Limoges University Hospital, Limoges
  - Nancy University Hospital, Nancy
  - Nantes University Hospital, Nantes
  - Lariboisière University Hospital (AP-HP), Paris
  - La Pitié-Salpétrière University Hospital (AP-HP), Paris
  - Sainte Anne Hospital, Paris
  - Rotschild Fundation, Paris
  - Poitiers University Hospital, Poitiers
  - Rennes University Hospital, Rennes
  - Rouen University Hospital, Rouen
  - Toulouse University Hospital, Toulouse
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] L'Allinec V, Chatel S, Karakachoff M, Bourcereau E, Lamoureux Z, Gaignard A, Autrusseau F, Jouan S, Vion AC, Loirand G, Desal H, Naggara O, Redon R, Edjlali M, Bourcier R. Prediction of Unruptured Intracranial Aneurysm Evolution: The UCAN Project. Neurosurgery. 2020 Jul 1;87(1):150-156. doi: 10.1093/neuros/nyaa093. PMID 32374868